CLINICAL TRIAL: NCT01154231
Title: BENEFIX(REGISTERED) INTRAVENOUS 500 1000 2000 DRUG USE RESULTS SURVEY (ALL-CASE SURVEILLANCE)
Brief Title: BeneFIX Drug Use Results Survey [All-Case Surveillance]
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3090X1-4415; B1821009 (Other: Alias Study Number)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia B
Keywords: BeneFIX Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nonacog Alfa (Genetical Recombination)
  Interventions: Drug: Nonacog Alfa (Genetical Recombination)

INTERVENTIONS:
Drug: Nonacog Alfa (Genetical Recombination) — Patients with hemophilia B (congenital blood coagulation factor IX deficiency) who are administered this drug.
  Patients with hemophilia B are either patients for whom treatment was already started with a blood coagulation factor IX product ("Previously treated patients": hereinafter, "PTPs") or patients who have no history of treatment with a blood coagulation factor IX product in the past and for whom treatment will be started with this drug for the first time ("Previously untreated patients": hereinafter, "PUPs").
  The definition of PUPs in this survey is "Patients in whom the total number of days of administration of a blood coagulation factor IX product other than this drug before administration of this drug was 3 exposure days (actual number of days of administration: hereinafter, "EDs") or less."
  Other Names: BeneFIX

SUMMARY:
The survey is intended to investigate the following matters, etc. under the actual use status after marketing in all patients who are administered this drug for a certain period of time after the launch.

1. Occurrence status of adverse events
2. Factors that may influence the safety
3. Efficacy In addition, the following occurrence statuses will be investigated as priority items of the survey: Incidence rate of inhibitor, reduction in drug, efficacy, Allergic reaction, and Thrombosis.

DETAILED DESCRIPTION:
Patients with hemophilia B (congenital blood coagulation factor IX deficiency) who are administered this drug.

Patients with hemophilia B are either patients for whom treatment was already started with a blood coagulation factor IX product ("Previously treated patients": hereinafter, "PTPs") or patients who have no history of treatment with a blood coagulation factor IX product in the past and for whom treatment will be started with this drug for the first time ("Previously untreated patients": hereinafter, "PUPs").

The definition of PUPs in this survey is "Patients in whom the total number of days of administration of a blood coagulation factor IX product other than this drug before administration of this drug was 3 exposure days (actual number of days of administration: hereinafter, "EDs") or less."

ELIGIBILITY:
Inclusion Criteria:

* All patients with hemophilia B scheduled to receive treatment with BeneFIX will be eligible for the surveillance.
* No patient will be excluded because of prior inhibitor history; however, complete patient history and demographics will be collected.

Exclusion Criteria:

* Patients not administered BeneFIX.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia B (congenital blood coagulation factor IX deficiency) who are administered this drug.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2014-08-29 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Tokyo Medical University Hospital, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090X1-4415&StudyName=BeneFIX%20Drug%20Use%20Results%20Survey%20%5BAll-Case%20Surveillance%5D

RESULTS

PARTICIPANT FLOW:
Groups:
- BeneFIX (Nonacog Alfa): Participants, who received BeneFIX injection intravenously as indicated in the approved local product document, were observed for periods of 1 year for PTPs and 2 years for PUPs. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | BeneFIX (Nonacog Alfa)
Started | 314
Completed | 312
Not Completed | 2
Not completed — Safety Unassessable, No Drug Admin. | 1
Not completed — No Info. After 1st Day, No Drug Admin. | 1

BASELINE CHARACTERISTICS:
Population: A total of 314 participants completed the study. Of the 314 participants, 2 participants were excluded from the baseline analysis. One was excluded due to no information after first day of treatment and no drug administration, the other due to safety not assessable and no drug administration.
Arm/Group | BeneFIX (Nonacog Alfa)
Number analyzed (Participants) | 312
Age, Customized [Number; unit: Participants]
  <15 years | 124
  ≥15 years <65 years | 179
  ≥65 years | 8
  Unknown | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 308
Previously Treated History [Number; unit: Participants] — PTPs refer to previously treated patients. PUPs refer to previously untreated patients.
  Participants
    PTPs | 281
    PUPs | 28
    Others | 3
Severity [Number; unit: Participans] — The severity of heamophilia B was defined as follows; severe, blood coagulation factor IX activity less than 1%; moderate, 1% to 5%; mild, more than 1%.
  Participans
    Severe | 156
    Moderate | 98
    Mild | 43
    Unknown | 15
Number of Bleeding in the Past 1 Year [Number; unit: Participants]
  ˂10 Times | 194
  ≥10 to ˂50 Times | 73
  ≥50 Times | 8
  Unknown | 37
History of Inhibitor [Number; unit: Participants]
  Yes | 6
  No | 306
Hemophilic Arthropathy [Number; unit: Participants]
  Yes | 133
  No | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Episodes (Annual Bleeding Event Rate) During Periodic Replacement Therapy
Description: Annual bleeding rate (ABR) was calculated as the number of total bleeding events occured during prophylaxis period devided by the period (events/year). ABR for other replacement treatment period was also calculated to evaluate the differences between types of treatment. If the period used for ABR calculation was less or equal than 7 days, the relevant data was regarded as missing.
Time Frame: 2 years for PTPs, 1 year for PUPs
Population: Efficacy analysis set who recieved at least one administration and had at least one efficacy evaluation was used for this analysis.
Measure: Median (Inter-Quartile Range); unit: Bleeding events/year
Arm/Group | BeneFIX (Nonacog Alfa)
Number analyzed (Participants) | 178
Bleeding events/year | 2.00 (11.29) [0.00 to 5.99]

2. Primary Outcome: Number of Administrations Required for Hemostasis for Bleeding Events
Description: Mean number of administrations for hemostasis in replacement therapy for bleeding events.
Time Frame: 2 years for PTPs, 1 year for PUPs
Population: as for outcome 1
Measure: Mean (Full Range); unit: administrations
Units Other Than Participants: dosing for hemostasis
Arm/Group | BeneFIX (Nonacog Alfa)
Number analyzed (Participants) | 112
Number analyzed (dosing for hemostasis) | 1161
administrations | 1.8 (4.18) [0.31 to 33]

3. Secondary Outcome: Subjective Evaluation of Each Therapeutic Administration for Bleeding Episodes
Description: Propotion of subjects whose physicians evaluated the effect of BeneFIX for bleeding episodes as excellent or good was calculated.
Time Frame: 2 years for PTPs, 1 year for PUPs
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: evaluations by physicians
Arm/Group | BeneFIX (Nonacog Alfa)
Number analyzed (Participants) | 112
Number analyzed (evaluations by physicians) | 671
percentage | 93.7 [91.6 to 95.5]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | BeneFIX (Nonacog Alfa)
Serious Adverse Events (participants affected / at risk) | 5/312
Other Adverse Events (participants affected / at risk) | 35/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (Nonacog Alfa) (N=312)
Herpes zoster (Infections and infestations) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Pulmonary artery atresia (Congenital, familial and genetic disorders) | 1
Gait disturbance (General disorders) | 1
Anti factor IX antibody positive (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (Nonacog Alfa) (N=312)
Nasopharyngitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Adenovirus infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Injection site pruritus (General disorders) | 1
Pyrexia (General disorders) | 1
CD4 lymphocytes decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.